CLINICAL TRIAL: NCT05196815
Title: Utility of Novel Echocardiographic and Invasive Haemodynamic Measurements in the Assessment of Patients Low Flow Low Gradient Aortic Stenosis Undergoing TAVI
Brief Title: Novel Echocardiographic and Invasive Haemodynamic Measurements in the Assessment of Patients Low Flow Low Gradient Aortic Stenosis Undergoing TAVI
Acronym: LFLG
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The Royal Wolverhampton Hospitals NHS Trust (Other Government)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2021CAR121
Record Dates: First submitted 2021-12-14; First posted 2022-01-19 (Actual); Last update posted 2025-01-06 (Actual); Status verified 2025-01

CONDITIONS: Cardiovascular Abnormalities
MeSH Terms: conditions — Cardiovascular Abnormalities | interventions — High-Energy Shock Waves; Catheters; X-Rays; Dobutamine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- The Royal Wolverhampton NHS Trust- New Cross Hospital (Experimental)
  Interventions: Other: Ultrasound; Procedure: Catheters; Procedure: Soft study wire; Radiation: X-ray; Drug: Dobutamine

INTERVENTIONS:
Other: Ultrasound — Participants will have a routine ultrasound of the heart (echocardiogram) before the procedure. During this test we will take a few extra measurements, this will not add any significant time to the scan
Procedure: Catheters — During the TAVI procedure 3 catheters (tubes) will be inserted into the blood vessels at the top of the participants legs as per normal standard care (there will be no extra skin punctures as part of the study).
Procedure: Soft study wire — Participants will have a soft study wire inserted to measure the pressure in the left ventricle. This step is in addition to standard care.
Radiation: X-ray — Participants will have chests x-ray when the soft study wire is inserted.
Drug: Dobutamine — Participants will be given a low dose infusion of dobutamine, to make the heart pump quicker and more vigorously.. This will last for approximately 5 minutes

SUMMARY:
In this study the investigators will assess a variety of novel markers of heart strength (contractility) and assess whether they can give a clearer indication of how well patients with weak hearts respond to the TAVI procedure.

The investigators will perform a stress echocardiogram prior to each TAVI procedure and measure the global longitudinal strain (GLS) in the left ventricle (LV) heart muscle, a detailed marker of muscle strength.

The investigators will then proceed to the TAVI procedure and measure the contractility of the main pumping chamber in the heart before and after giving a very low dose of an adrenaline -like drug (dobutamine). The patient will already have received this short acting drug (at the same and higher doses) during their routine care planning stress echocardiogram.

DETAILED DESCRIPTION:
In this study the investigators will assess a variety of novel markers of heart strength (contractility) and assess whether they can give a clearer indication of how well patients with weak hearts respond to the TAVI procedure.

The investigators will perform a stress echocardiogram prior to each TAVI procedure and measure the global longitudinal strain (GLS) in the left ventricle (LV) heart muscle, a detailed marker of muscle strength.

The investigators will then proceed to the TAVI procedure and measure the contractility of the main pumping chamber in the heart before and after giving a very low dose of an adrenaline -like drug (dobutamine). The patient will already have received this short acting drug (at the same and higher doses) during their routine care planning stress echocardiogram.

The investigators will also measure the pressure across the aortic valve, known as the trans-aortic gradient, using the pressure wire (PW) and a standard (multipurpose) heart catheter. The investigators will repeat the resting measures (i.e. without pacing or dobutamine) at the end of the procedure to measure the early change in left ventricular contractility and then repeat the echocardiogram immediately and after 3 months to assess the outcome of the TAVI procedure in terms of left ventricular function volume and function

ELIGIBILITY:
Inclusion Criteria:

1. Patients presenting symptomatic AS listed for TAVI
2. Native aortic valve disease
3. Ejection fraction </= 40%
4. Mean trans aortic gradient (echo) of <35 mmHg
5. AVA </= 1cm2
6. Able to give written informed consent prior to enrolment in the study
7. No contraindication to study procedures
8. CT scan confirmed severe AS
9. *Able and willing to return to the implanting site for the follow-up visits*

Exclusion Criteria:

1. Unable to provide formal written consent
2. Known pseudo-severe AS prior to TAVI
3. Known allergy to agents required for stress echocardiography
4. Known hypersensitivity or contraindication to aspirin, heparin, clopidogrel, Nitinol, or sensitivity to contrast media, which cannot be adequately premedicated. *
5. Any clinical contraindication to TAVI procedure

This pilot study will be restricted to English speaking subjects.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 7 (Actual)
Dates: Start 2022-07-01 (Actual); Primary Completion 2024-03-01 (Actual); Study Completion 2024-03-01 (Actual)

PRIMARY OUTCOMES:
Change in LV ejection fraction at 3 months compared to pre procedural readings. | 3 months
  Change in LV ejection fraction as a percentage
Change in LV Volume at 3 months compared to pre procedural readings. | 3 months
  Change in LV Volume measured by BSA, mL/m2
Change in global longitudinal strain at 3 months compared to pre procedural readings. | 3 months
  Change in global longitudinal strain measured by percentage
Change in fractional shortening by echocardiography at 3 months compared to pre procedural readings. | 3 months
  Change in fractional shortening measured by percentage
The change in contractility (dP/dT) with low dose dobutamine stress prior to TAVI, measured by invasive Pressure Wire | 3 months
  The change in contractility (dP/dT) with low dose dobutamine stress prior to TAVI, measured by invasive Pressure Wire
The change in aortic trans-valvular gradient with low dose dobutamine stress during TAVI prior to AV treatment. | 3 months
  The change in aortic trans-valvular gradient measured by mmHg
The change in contractility (dP/dT) from pre to post procedure at 3 months. | 3 months
  The change in derivative of pressure over time (dP/dT) is measured by the change in pressure per unit time. Measured ventricular pressure provides an indication of the contractility or relaxation of the ventricles of a heart. In this way, the derivative of pressure over time (dP/dt) provides a biphasic signal that can be used to evaluate acute directional changes of contractility

CONTACTS AND LOCATIONS:
Overall Officials: James Cotton, Principal Investigator — The Royal Wolverhampton NHS Trust
Locations (1):
- The Royal Wolverhampton NHS Trust, Wolverhampton, West Midlands, United Kingdom